CLINICAL TRIAL: NCT03825926
Title: Early Screening of Gestational Diabetes Mellitus and Prospective Cohort Study of Postpartum Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.CK.001
Record Dates: First submitted 2019-01-24; First posted 2019-02-01 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — whole blood and placenta, umbilical cord endothelial tissue and umbilical cord blood after the delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational Diabetes Mellitus: The diagnosis of GDM is based on a 75-g oral glucose tolerance test (OGTT) performed between 24 and 28 gestational weeks, according to the American diabetes association (ADA) criteria (fasting ≥ 5.1 mmol/L, 1 h ≥ 10.0 mmol/L, 2 h ≥ 8.5 mmol/L). Recruited patients were accepted the standard of treatment of GDM according to the American college of obstetricians and gynecologists (ACOG) practice bulletin on gestational diabetes mellitus.
- Non-Gestational Diabetes Mellitus: normal group

SUMMARY:
Extraction of whole blood from 10 to 15ml at 24 weeks before pregnancy test, with a view to early detection of GDM, provides evidence for early intervention to improve maternal pregnancy outcomes and metabolic abnormalities.

DETAILED DESCRIPTION:
1. Pregnancy cohort management and follow-up

1. All pregnant women in the group are included in the study queue and have a uniform number, which is followed up until the birth.
2. Detailed case reporting forms have been developed to record the data.
3. We have set up a relatively complete electronic database of obstetrics, which will include modules related to this study, which will be available for this project management data.
4. This project has a full-time research assistant as a high-grade nurse. He is responsible for the maternity examination and follow-up of pregnant women in the group and ensures the norms of the maternity inspection process so as to reduce the heterogeneity caused by inconsistent labor inspection times. All birth tests are conducted in accordance with the Guidelines for Pre-conception and Pregnancy Care.
5. Pregnant women diagnosed as GDM will be managed in accordance with the Guide for the Diagnosis and Treatment of Pregnancy Combined with Diabetes(2014).
6. In addition to conducting five blood samples and tissue collection, we have followed the existing clinical principles and guidelines in handling and intervening in pregnancy and childbirth-related issues.

2. Collection Time and Content of Clinical Indicators

1. Data collection time nodes: pregnancy 11-13 + 6 weeks, pregnancy 18-20 weeks, pregnancy 24-28 weeks, hospitalization during childbirth, six months after delivery.
2. When entering the group: age, pre-pregnancy weight, height, pregnancy, birth; Ask for history, history of marriage and family history in detail.
3. items to be collected for each birth test: weight, blood pressure, palace height, abdominal circumference; Assess complications during pregnancy.
4. Pregnancy B Super monitoring: At least 11-13 weeks of early pregnancy B super, 18-24 weeks of three-dimensional color super, 32 weeks and 37 weeks of color Super.

3. Collection time and content of laboratory indicators

1. Data collection time nodes: pregnancy 11-13 + 6 weeks, pregnancy 18-20 weeks, pregnancy 24-28 weeks, hospitalization during childbirth, six months after delivery.
2. When entering the group(11-13 + 6 weeks of pregnancy): Extraction of blood 10 ~ 15ml to detect relevant metabolic biological indicators in the molecular influence center laboratory of our hospital or the National University of China Gene Company, such as: Asprosin, leptin, etc..
3. Pregnancy 18-20 weeks ago: Extraction of blood 10 ~ 15ml in our laboratory molecular center laboratory to detect related metabolic biological indicators, such as: Asprosin, leptin and so on.
4. Pregnancy 24-28 weeks: draw blood 10 ~ 15ml. Routine clinical examination and examination of OGTT test in our hospital examination department, and the detection of blood lipid and glycosylated hemoglobin. Additional metabolic biomarkers are detected in the central laboratory of molecular in our hospital.
5. Inpatient delivery: routine inpatient blood collection examination, and blood extraction 10 ~ 15ml in our hospital molecular influence center laboratory to detect related metabolic biological indicators, such as: Asprosin, leptin and so on.
6. Six months after delivery: GDM group patients will undergo postpartum review in our hospital, draw blood 10 ~ 15ml in our hospital molecular influence center laboratory to detect related metabolic biological indicators, such as: Asprosin, leptin, etc..

4. GDM diagnostic criteria 75g OGTT method: OGTT fasting at least 8 hours before the test, continuous 3 days normal diet before the test, that is, eating carbohydrates not less than 150g per day, sit-in during the examination, smoking ban. At the time of examination, 5 min was taken orally with a liquid of 75g of glucose, and 1 and 2 hours of venous blood(calculated from the start of drinking glucose water) was extracted from the pregnant woman before and after taking sugar, and placed in a test tube containing sodium fluoride. Glucose oxidase method was used to determine blood sugar level.

The diagnostic criteria for 75g OGTT: 1, 2 H before and after taking sugar, 3 blood sugar values should be below 5.1, 10.0, 8.5 mmol/L(92, 180, 153 mg/dl), respectively. Any blood sugar value that reaches or exceeds the above criteria is diagnosed as GDM.

5. Measures to manage GDM Since there is currently no basis for the GDM management of pregnant women who meet the GDM diagnostic criteria 24 weeks ago, the OGTT anomaly is sufficient to diagnose the GDM for the standardized management of gestational diabetes. Refer specifically to the Guide for the Diagnosis and Treatment of Pregnancy with Diabetes(2014). Any test of abnormal glycolipids metabolism, or any other test to diagnose diabetes complicated pregnancy(this diagnosis is different from GDM, with an empty abdomen of 7.0 mmol/L or 2 H to 11.1 mmol/L), Both began management of diabetes during pregnancy(the group will withdraw from the study).

6. Monitoring and follow-up during childbirth. 6.1 Clinical data collection on pregnant women during childbirth Items to be collected during the birth of a pregnant woman: pregnancy, perinatal complications, mode of delivery, and the duration of the birth.

6.2 Laboratory data collection on pregnant women during childbirth Pregnant women during childbirth: peripheral blood sugar test(fasting and 2 hours after meal blood sugar), glycated hemoglobin.

6.3 Neonatal clinical and laboratory data collection

1. The items to be collected by newborns: birth weight, length, head circumference, shoulder circumference, abdominal circumference, upper arm circumference, birth style, newborn Apgar score, whether to transfer to Neonatal Intensive Care Unit, Neonatal complications(hypoglycemia, neonatal hypocalcemia, neonatal hyperbilirubinemia, neonatal erythrocytosis, neonatal asphyxia, neonatal respiratory distress syndrome, etc..)
2. Neonatal test: umbilical blood sugar(GDM group only)

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-40 years old. The age is determined by the date of birth and the expected date of birth of the identity card.
2. Age of entry into the group: Before 16 weeks of pregnancy. The determination of pregnancy week refers to the Hyperglycemia and Adverse Pregnancy Outcomes research report method. Specifically, first, if the pregnant woman's menstruation is regular, the pregnancy week is calculated according to the last menstrual time. If the menstruation is irregular or the last period can not be determined, the pregnancy week is calculated using B-ultrasound results during the period of 6-24 weeks. Second, if menstruation is regular, but there is a large difference with the B-super estimated expected date of delivery, it is more than 5 days different from the 6-13 weeks B-super result, or more than 10 days different from the 14-24 weeks result, still correcting the pregnancy week according to the B-super result.
3. Number of pregnancies: This study does not limit the number of pregnancies. In order to improve consistency and compare with previous studies, all those who entered the group were single pregnancies.
4. Prenatal examination: In order to improve the consistency of the study, the patients in the group were all examined regularly in our hospital, and the important laboratory results accepted by the research institute were all conducted in our hospital.

Exclusion Criteria:

1. Pregnancy week: At the time of the visit, the pregnancy week has exceeded 24 weeks, or the pregnancy week can not be determined.
2. Pregnancy mode: unnatural pregnancy(including ovulatory drugs, test-tube infants, etc.).
3. Diabetes combined with pregnancy: previously diagnosed diabetes; Or early pregnancy fasting blood sugar ≥ 7.0 mmol/L and diagnosed diabetes combined pregnancy; Or by other situations(random blood sugar > 11.1 mmol/L with diabetes symptoms) Diagnosis of diabetes combined with pregnancy.
4. As a result of the combination of other diseases, drugs that affect glucose metabolism, such as glucocorticoids and diuretics, are being taken.
5. Combine other diseases that affect sugar metabolism, such as hyperthyroidism, history of polycystic ovary syndrome, etc..
6. Because the target population in this study is a normal population, people with high risk factors for GDM will be excluded: such as the family history of type 2 diabetes, the history of huge childbirth, the past pregnancy combined with GDM, and obesity(BMI≥30kg/m2), poor maternity history, etc..
7. Those who do not agree to draw blood before 24 weeks of pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: 1. Inform interviewees who meet the requirements for access of the relevant research content and risks, obtain their consent, and sign the informed consent.
  2. pregnant women during the birth test, pregnancy 11 ~ 13 + 6 weeks and pregnancy 18-20 weeks, respectively, 10 ~ 15ml.
  3. Clinical blood samples will also be recovered for scientific purposes during 24-28 weeks of routine delivery and prior to delivery in hospital.
  4, after the birth to obtain placental tissue, umbilical cord endothelial tissue and umbilical cord blood.
  5.Follow up study the prognosis of gestational diabetes.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
New biomarkers levels in different pregnant weeks | the basic point (11-13+6 weeks), 18-20 weeks as the first changed point, 24-28 weeks as the second changed point,delivery weeks as the first outcome point, 6 months after delivery as the second outcome point
  1. Collect time: We will collect our sample in different pregnant weeks such as 11-13+6 weeks as early pregnancy, 18-20 weeks as compared mid-pregnancy, 24-28 weeks as the criteria mid-pregnancy, delivery weeks as the first outcome and 6 months after delivery time as the second outcome. This will be helpful to evaluate the criteria and explore pregnant glycolipid metabolism at new sight.
  2. Sample details: we will collect maternal blood for different pregnant weeks, neonatal cord blood, umbilical cord endothelial tissue and placenta after sign informed consent. All maternal and neonatal sample will tested the first step of new biomarkers by quantitative analysis methods such as mass spectrometers, immunohistochemistry and enzyme linked immunosorbent assay and so on. we will explore the changed range on those new biomarkers during early-mid-late pregnancy.
Evaluation of new biomarkers on the criteria | the basic point (11-13+6 weeks), 18-20 weeks as the first changed point, 24-28 weeks as the second changed point,delivery weeks as the first outcome point, 6 months after delivery as the second outcome point
  New biomarker tests show how consistent with GDM from The International Association of Diabetes and Pregnancy Study Groups criteria. We will do some new biomarker tests such as plasma mannose Levels, retinol-binding protein 4 and angiopoietin-like protein 4 and so on. There are 30-40 types' new biomarkers which is proved that it is relative with glycolipid metabolism on recent studies during 5 years.
  Evaluate the risk and the correlation between new biomarker and maternal and neonatal clinical outcomes.
Evaluation of the postpartum recovery follow up GDM or non-GDM | 3 days after delivery by conduct of interviews;
  World Health Organization Quality of Life Scale (WHOQOL 100) to evaluate subjects is only in 2 weeks for the labour.（All instructions and details are followed by the website:https://www.who.int/mental_health/publications/whoqol/en/ , such as scale design and scores calculation）.
Edinburgh postpartum depression scale (EPDS) follow up GDM or non-GDM | 3days after delivery by conduct of interviews; 6 months after delivery by wechat app
  There are three models on postpartum depression:the mild postpartum depression is 10-12 scores;the moderate postpartum depression is 13-15 scores;the severe postpartum depression is over 16 scores. Meanwhile, the scale design and other instructions come from the article.（Cox, J., Holden, J., & Sagovsky, R. (1987). Detection of Postnatal Depression: Development of the 10-item Edinburgh Postnatal Depression Scale. British Journal of Psychiatry, 150(6), 782-786. doi:10.1192/bjp.150.6.782）

SECONDARY OUTCOMES:
Expenditure on health products and drugs before diagnosed GDM | before 13+6 weeks as the first time, before the diagnosis of GDM as the second time
  we collect the name, type and value of health product and drugs before before diagnosed GDM among our samples
Expenditure on GDM after the diagnosis | after 24-28weeks as the first time, after 28 weeks until before the delivery hospitalization as the second time, the delivery hospitalization as the third time
  we count number of hospitalization and collect fee of outpatient and hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojuan Su, postgraduate, Study Chair — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the Fifth Affiliated Hospital of Sun Yat-sen University of Gynaecology and Obstetrics, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
This study is a prospective, single blind and observational clinical study. In order to evaluate the long-term effects of GDM on blood sugar, the early screening of GDM was studied through the changes in metabolic levels between different gestation ages.